CLINICAL TRIAL: NCT02788682
Title: Association of Vitamin D Binding Protein Polymorphisms With Response to Therapy in Chronic Hepatitis C Egyptian Patients
Brief Title: Association of Vitamin D Binding Protein Polymorphisms With Response to HCV Therapy
Status: Completed | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmed Mohamed Sayed Kamel, Teaching Assistant, Cairo University
Other Study IDs: CL (770)
Record Dates: First submitted 2016-05-27; First posted 2016-06-02 (Estimated); Last update posted 2016-07-26 (Estimated); Status verified 2016-07

CONDITIONS: Chronic Hepatitis C
Keywords: VDBP; single nucleotide polymorphisms (SNPs); interferon based therapy; Egypt
MeSH Terms: conditions — Hepatitis C, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — EDTA blood
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Patients: WT+ Diplotype
  Interventions: Genetic: WT+ Diplotype
- Controls: WT- Diplotype

INTERVENTIONS:
Genetic: WT+ Diplotype — 3 or 4 vitamin D binding protein major alleles
  Groups: Patients

SUMMARY:
Introduction: Vitamin D binding protein (VDBP) is a potential modulator of immune response and is associated with clinical progression of many diseases. Our aim is to assess influence of baseline 25-hydroxyvitamin D levels and VDBP single nucleotide polymorphisms (SNPs), rs4588 (C>A) and rs7041 (G>T), on baseline clinical parameters and response to interferon based therapy in chronic Hepatitis C patients in Egypt.

Methodology: Genotyping will be performed by RFLP (Restriction Fragment Length Polymorphism) in treatment naïve Hepatitis C patients and healthy controls. Vitamin D levels will be assessed by ELISA. HCV RNA quantification will be performed by PCR to assess therapy outcome.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years and ≤ 60 years, fasting blood sugar less than 115 mg/dl or 20% upper normal limit (140 mg/dl), HBA1C ≤ 7.5% in diabetic patients, normal serum creatinine, normal thyroid stimulating hormone level, negative Hepatitis B surface antigen, hemoglobin ≥ 12g/dl for male or ≥ 11g/dl for female, total leukocytes ≥ 3,500/mm3, ANC ≥ 1500/mm3, platelets ≥ 100,000/mm3, presence of HCV RNA by PCR and elevated liver enzymes within the preceding 6 months for patients with F1 fibrosis stage.

Exclusion Criteria:

* hypersensitivity to interferon or ribavirin, decompensated liver cirrhosis (presence of ascites, esophageal varices or hepatic encephalopathy), hepatocellular carcinoma, body mass index>35 Kg/m2 and vitamin D supplementation.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Chronic Hepatitis C patients in Egypt
Sampling Method: Non-Probability Sample
Enrollment: 162 (Actual)
Dates: Start 2013-09; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
SVR | 72 weeks

IPD SHARING:
Plan to Share IPD: No